CLINICAL TRIAL: NCT06503276
Title: The Efficacy of Combination of Orelabrutinib and Ultra-low Dose Radiotherapy in the First-line Treatment of Early Ocular Adnexal Extranodal Marginal Zone B-cell Lymphoma
Brief Title: The Treatment of Ocular Adnexal Extranodal Marginal Zone B-cell Lymphoma by Orelabrutinib and Radiotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Jun Shi, Hematology Department Director, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OA-EMZL-1
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Extranodal Marginal Zone B-cell Lymphoma
MeSH Terms: interventions — orelabrutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orelabrutinib+Ultra-low dose radiotherapy (Experimental): Patients will receive radiotherapy 2Gy twice and orelabrutinib orally for 4 months, 150mg Qd
  Interventions: Drug: Orelabrutinib; Radiation: Ultra-low dose radiotherapy

INTERVENTIONS:
Drug: Orelabrutinib — Orelabrutinib PO will be administered as per the schedule specified in the respective arm
Radiation: Ultra-low dose radiotherapy — 2 Gy radiotherapy will be administerd twice in the first cycle

SUMMARY:
Extranodal marginal zone B-cell lymphoma (EMZL) is the most common lymphoma of the ocular adnexa (OA), accounting for approximately 60%. As a special part of the body, there is no consensus on the optimal treatment strategy for OA-EMZL. Studies have shown that patients who wait for postoperative observation have a 5-year PFS of approximately 80% and a 10-year PFS of 63%. Therefore, radiotherapy remains an important treatment for stage I/II OA-EMZL patients, but the dosage of radiotherapy remains controversial. In 2014, Hoskin PJ et al. found that the complete response rate and effective rate of patients in the standard 24Gy radiation dose group were 71% and 91%, while those in the 4Gy radiation dose group were 55% and 87%, respectively. Meanwhile, the PFS of patients with 4Gy radiation dose was lower than that of the group with 24Gy radiation dose, but there was no significant difference in OS between the two groups. However, in a study conducted by Chelius M et al. in 2021, they found that the incidence of both early and late toxic effects was significantly higher in the>4Gy radiation dose group than in the<4Gy radiation dose group. These toxic effects inevitably affect the quality of life of patients. Therefore, investigators plan to adopt a combination of ultra-low dose radiotherapy and drug therapy, which not only reduces the side effects of radiotherapy, but also improves the complete response rate of treatment and reduces disease progression or recurrence. However, studies have shown that radiotherapy combined with rituximab cannot improve the disease-specific survival rate of OA-EMZL. Therefore, BTK inhibitors (BTKi), as a novel targeted drug for the treatment of EMZL, have been used to treat relapsed and refractory EZML by interfering with BCR signals. Based on the above research, investigators plan to explore the efficacy of combination therapy with Orelabrutinib and ultra-low dose radiotherapy (4Gy) in the treatment of stage I/II OA-EMZL.

ELIGIBILITY:
Inclusion Criteria:

* 1: Male or female, aged 18-75 years.

  2: Newly diagnosed patients with Marginal Zone B-cell lymphoma of ocular adnexa confirmed by surgical biopsy, with early Ann Arbor stage (stage I/II) and evaluable lesions (> 1cm) on imaging.

  3: Laboratory tests prior to admission must meet the following criteria: white blood cell count ≥3.0x10^9/L, absolute neutrophil count ≥1.5 x10^9/L, hemoglobin ≥90g /L, platelets ≥75x 10^9/L.

Liver function: transaminase levels≤3 times the upper limit of normal, bilirubin levels ≤1.5 times the upper limit of normal.

Serum creatinine clearance ≥30 mL/min. Myocardial enzymes < 2 times the upper limit of normal (same age). ECOG score 0-2.

4: All subjects must provide informed consent and voluntarily sign the written informed consent form themselves or through their legal representatives before participating in the study.

Exclusion Criteria:

* 1: Pregnant or lactating women, and women of childbearing potential who refuse to use contraceptive measures.

  2: Inability to swallow, chronic diarrhea, or intestinal obstruction, or any condition that affects drug use and absorption.

  3: Pre-trial treatment: Use of drugs that significantly affect the P450 metabolic enzyme pathway within 2 weeks before the screening period.

Current use of cyclosporins or fibrates. Participation in other clinical studies and use of investigational drugs within 28 days prior to the initiation of the study drug.

The need to use concomitant drugs that may prolong QTc or induce tip torsion ventricular TdP, in addition to antimicrobials used as standard care to prevent or treat infections and other such drugs that investigators consider essential for treatment.

4: Evidence of current uncontrolled cardiovascular disease, including: Uncontrolled high blood pressure. Uncontrolled arrhythmia. Symptomatic congestive heart failure. Unstable angina. Myocardial infarction within the past 6 months. Severe acute or chronic infections requiring systemic treatment. Known human immunodeficiency virus (HIV) infection , or active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.

Have a history of uncontrolled seizures, a central nervous system disorder, or a mental illness.

5: History of malignant tumors other than OA-EMZL, unless the patient has been cured for more than 3 years.

6: Any past or current disease, treatment, or laboratory abnormality that may interfere with the study results or affect the subject's full participation in the study, or the investigator deems the subject unfit to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate | End of treatment (4 months after administration)
  Percentage of participants with complete response was determined on the basis of investigator assessments

CONTACTS AND LOCATIONS:
Overall Officials: Jun Shi, Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China